CLINICAL TRIAL: NCT00121823
Title: Malaria Infection Diagnosed by PCR as a Means of Evaluating Pre-erythrocytic Candidate Malaria Vaccines
Brief Title: Malaria Infection Diagnosed by Polymerase Chain Reaction (PCR) as a Means of Evaluating Pre-erythrocytic Candidate Malaria Vaccines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); University of Oxford (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: ITDCVG37; VAC 029
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Malaria; PCR; Vaccines; Acceptability
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Biological: FP9 ME-TRAP
Biological: MVA ME-TRAP

SUMMARY:
The ability to test candidate pre-erythrocytic stage malaria vaccines, using a well-established sporozoite challenge model, in a field setting with group sizes of tens rather than hundreds of volunteers would greatly facilitate identification of the most promising vaccine candidates. The investigators assessed the suitability and acceptability of this method in a field trial in semi-immune volunteers exposed to natural infection during the high malaria transmission season.

DETAILED DESCRIPTION:
Objective

The primary objective of the study was to determine if the very sensitive PCR technique, capable of detecting malaria parasites at low densities could be used as an economical method of undertaking preliminary field evaluation of pre-erythrocytic malaria vaccines. A secondary objective was to determine if the intensive blood sampling that this method requires would be acceptable.

Study area

This study was conducted from June to October 2004 when the incidence of malaria in The Gambia is highest. Volunteers were recruited from 9 villages east of Farafenni, a town which is 200km east of the capital city, Banjul. Malaria is highly seasonal in this area with an entomological inoculation rate between 10 and 50 infectious bites per year.

Study population

Healthy volunteers aged between 15-45 years were screened at two centres for their eligibility to take part in the study. Screening involved a thorough physical examination as well as blood sampling tests for haematological (full blood count, packed cell volume [PCV]), renal (plasma creatinine level) and hepatic (alanine amino transferase) tests and for HIV 1 and 2 tests by ELISA. A glucose-6-phosphate dehydrogenase (G6PD) deficiency test was carried out because of the risk involved with administering the study drugs Primaquine and Lapdap to volunteers who are G6PD deficient. Exclusion criteria included a PCV < 30%, raised plasma creatinine (> 130 micromoles/litre) or ALT levels (> 42 IU/litre), G6PD deficiency, simultaneous participation in another clinical trial, blood transfusion in the month prior to vaccination, previous experimental malaria vaccination, administration of another vaccine within 2 weeks of vaccination, allergy to any previous vaccination or to sulphadoxine/pyrimethamine, history of splenectomy and any treatment with immunosuppressive drugs.

Study procedure

Eligible volunteers were enrolled into the study after written, informed consent was obtained. All eligible volunteers were issued a unique number and a photo identification card. Volunteers were randomly allocated into three groups to receive either two 5 x10^7 pfu doses of FP9 ME-TRAP followed by a single dose of 1 x 10^8 pfu MVA ME-TRAP (malaria vaccine group) or 3 doses of rabies vaccine (Fansidar and rabies groups). All vaccines were give 4 weeks apart and were administered intradermally. Following vaccination, all volunteers were observed for 1 hr and given a course of anti-pyretic (paracetamol) to take if required. In addition, home visits were made by field workers on days 1, 2, 7 and 28 after each vaccination to record adverse events using a standard diary card. All volunteers received a single dose of Primaquine (30mg) 7 days before the final dose of vaccination as radical cure for gametocytes and a 3-day course of the short acting anti-malaria drugs, Lapdap and Artesunate in combination starting on the day of final vaccination to clear any asexual forms of the parasite before the follow-up period. Additionally, volunteers in the Fansidar group received the long acting anti-malarial drug and were expected to remain PCR negative throughout the follow-up period. Volunteers were followed up intensively for 28 days starting 7days after the last vaccination. The period of follow-up was timed to correspond with the period of high malaria transmission. Follow-up was by daily finger-pricks to obtain 0.5mls of blood in a microtainer for PCR analysis and a duplicate blood film for estimation of malaria parasites. Laboratory staff that conducted immunoassays and PCR analysis were blind to the group allocation of volunteers until after approval of the analysis plan by the Data Safety Monitoring Board (DSMB).

Sample size

Based on practical and statistical considerations the researchers proposed to enroll 40 volunteers per group (a total of 120). Allowing for a steady rate of drop-out during follow up amounting to total of 20% of subjects by the end of the trial, the trial has at least 80% power to detect a difference in time to infection between the malaria vaccine and rabies groups, if the vaccine efficacy is at least 60%, and at least 70% of the control group volunteers develop detected parasitaemia during the trial.

Data Safety Monitoring Board (DSMB)

A DSMB was set up to oversee the conduct of the trial and approve the analytical plan before unblinding the laboratory staff. The trial was conducted according to ICH Good Clinical Practice guidelines and was guided by the Medical Research Council regulations for the conduct of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 15-45 years
* Signed informed consent form

Exclusion Criteria:

* Clinically significant history of skin disorder (eczema, psoriasis, etc.), allergy, immunodeficiency, cardiovascular disease, respiratory disease, endocrine disorder, liver disease, renal disease, gastrointestinal disease or neurological illness.
* Any clinical evidence of immunosuppression such as oral candida, stomatitis, aphthous or septic ulceration, septic skin lesions or any clinical or laboratory evidence of infection or immunosuppression.
* History of splenectomy
* Haematocrit of less than 30%
* Serum creatinine concentration >130mmol/L
* Serum ALT concentration >80 IU/L
* Blood transfusion within one month of the beginning of the study
* History of vaccination with a previous experimental malaria vaccine
* Administration of any other vaccine or immunoglobulin within two weeks of scheduled vaccination.
* Positive HIV antibody test.
* Positive colorimetric test for G-6-P-D deficiency.
* Current participation in another clinical trial, or within 12 weeks of this study.
* Lack of parental consent if volunteer is aged under 18
* Likelihood of travel away from the study area for the duration of the study
* Any other finding which in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial
* Known allergy to sulfadoxine/pyrimethamine (SP), Artesunate or Lapdap
* Drug or alcohol addiction
* Egg allergy

Ages: 15 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 2004-06; Study Completion 2004-12

PRIMARY OUTCOMES:
Suitability and acceptability of study method

SECONDARY OUTCOMES:
Prevention of malaria parasitaemia

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, Phd, Study Chair — University of Oxford; Brian M Greenwood, MD, Study Director — Gates Malaria Partnership
Locations (1):
- Medical Research Council Laboratories, Banjul, The Gambia